CLINICAL TRIAL: NCT04194983
Title: To Examine the Effect of Dietary Supplementation With Fish Oils With Dairy or Plant Based Lipids on Mitochondrial, Physical, and Cognitive Function, in Elderly Humans
Brief Title: The Effect of Fish Oils With Dairy or Plant Based Lipids on Mitochondrial and Physical, and Cognitive Function, in Elderly Humans
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to COVID-19 and lack of financial means to continue
Sponsor: Maastricht University (Other)
Collaborators: Wageningen University and Research (Other); Netherlands Organisation for Scientific Research (Other Government); Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL68966.068.19
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Ageing; Mitochondrial Function; Physical Function; Cognitive Function
Keywords: Ageing; Mitochondrial Function; Physical Function; Cognitive Function; Dietary Fat
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Intervention Model Description: A multicenter, double-blind, randomised, controlled, parallel trial, where fish oils combined with dairy or plant based fat supplements are consumed for 12-weeks.
Who Masked: Participant, Investigator
Masking Description: After subjects have successfully completed the screening, they will be randomly allocated in a 1:1 ratio, using a 4-code system, to one of the two interventions (intervention or control). The intervention and control will each be individually coded with a randomly generated 3 letter coding system with 2 codes allocated to intervention product and the other 2 codes allocated to the control product. sachets will be generated by the product manufacturer and the corresponding blinding label will be added to the sachets, prior to shipment to the study sites. The un-blinding-key will be sent to the project leaders in sealed envelopes. In this way, both the participants and principle investigator will be blinded throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fish oils and dairy fats (Experimental)
  Interventions: Dietary Supplement: Fish oils and dairy fat
- Fish oils and plant fats (Placebo Comparator)
  Interventions: Dietary Supplement: Fish oils and plant fat

INTERVENTIONS:
Dietary Supplement: Fish oils and dairy fat — 12-weeks, 3x per day
  Arms: Fish oils and dairy fats
Dietary Supplement: Fish oils and plant fat — 12-weeks, 3x per day
  Arms: Fish oils and plant fats

SUMMARY:
The aim of this study is to determine whether dairy or plant based fats combined with fish oils can alter skeletal muscle mitochondrial, physical, and cognitive function.

DETAILED DESCRIPTION:
Physical and cognitive function decline as we get older and this may be due to changes within the mitochondria, organelles that regulate energy production in our cells. The ability of the mitochondria to produce energy can be affected by diet, and the composition of lipids in the cell is an important factor in determining how effective our mitochondria are. Dairy and plant based lipids differ in composition and therefore may differ in their ability to affect mitochondrial function when combined with fish oils (FO). The primary objective of this study is to determine whether supplementation with dairy or plant based fats combined with fish oils can alter skeletal muscle mitochondrial function. Additional exploratory objectives are 1) skeletal muscle and physical function and 2) cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Male or/and female;
* Caucasian;
* Age ≥ 65 years;
* BMI ≥ 20 kg/m2 ≤ 30 kg/m2;
* Normal physical activity levels: maximum of 1 hour per week engagement in structured exercise of moderate to high intensity;
* Subject should be in sufficient health to participate in the experiments, to be judged by the site-specific responsible physician, based on the subject's medical history.

Exclusion Criteria:

* Habitual smoker within the past 5 years;
* Excessive alcohol use (greater than 20g per day) and/or drug abuse;
* Subjects with diagnosed diabetes mellitus type 2;
* Significant food allergies or intolerances concerning the study products, e.g. cow's milk protein allergy
* Participation in another biomedical study possibly interfering with the study results within 1 month before the first study visit;
* Medication use e.g. antithrombotic medications known to hamper subject's safety during the study procedures;
* Subjects habitually taking fish oil supplements within 3-months of the initial study visit or habitually taking supplements that are likely to affect the main study outcomes;
* Subjects who do not want to be informed about unexpected medical findings;
* Subjects who do not want their treating physician to be informed about unexpected medical findings;
* Inability to participate and/or complete the required measurements

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Mitochondrial respiration | 12 weeks
  Ex vivo mitochondrial respiration expressed by O2flux in pmol/mg wet weight/second

SECONDARY OUTCOMES:
Physical function | 12 weeks
  Short physical Performance Battery (SPPB)
Cognitive Function | 12 Weeks
  Cambridge Neuropsychological Test Automated Battery (CANTAB)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, PhD, Principal Investigator — Maastricht University
Locations (2):
- Netherlands (2):
  - Wageningen University and Research, Wageningen, Gelderland
  - Maastricht University, Maastricht, Limburg